CLINICAL TRIAL: NCT01186601
Title: Open-label Study for an Exploration of Tumor Accumulation of the 18F Labeled PET/CT (Positron Emission Tomography / Computed Tomography) Tracer BAY94-9392 Following a Single Intravenous Administration of 300 MBq (Corresponding to </= 0.1 mg Total Quantity) in Patients With Prostate Cancer or Other Malignant Tumors
Brief Title: Exploration of Tumor Accumulation of BAY94-9392 in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15329
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasms
Keywords: Prostatic Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Melanoma; Neoplasm Metastasis
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: PET tracer (BAY94-9392)

INTERVENTIONS:
Drug: PET tracer (BAY94-9392) — A radioactive dose of 300 MBq of the study drug with a total quantity of </= 0.1 mg will be administered as slow intravenous bolus injection over up to 60 seconds

SUMMARY:
The study will be conducted as an open label, single-dose, explorative study with patients with histologically proven cancer and, preferably, tumor positive lesions in previously performed nuclear medicine imaging examinations.

The investigational drug will be given as a single administration in a dose of </= 0.1 mg BAY94-9392 (300 MBq, +/- 10%). The total duration of the study for each patient will be approximately 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Males/females >/= 18 years
* Patients with a diagnosis of primary prostate cancer (biopsy proven) and scheduled for radical prostatectomy or patients with prostate tumor recurrence (Patients with advanced tumor disease and a high likelihood to display lymph node metastasis are to be preferably included.)
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2, determined within one week prior to treatment with BAY94-9392
* Patient had an [18F]-fluorodeoxyglucose (FDG) PET/CT for detection, or staging, or restaging, or therapy response assessment that still showed tumor mass with high certainty for a cancer such as melanoma, or colorectal cancer, or head & neck cancer for which FDG-PET/CT is used in clinical routine, and the primary cancer disease is histologically confirmed. In case of recurrent disease confirmation of the primary tumor is sufficient
* No clinically relevant deviations in renal function as determined by Cockcroft and Gault method using serum creatinine at screening.

Exclusion Criteria:

* Concurrent severe and/or uncontrolled and/or unstable medical disease other than cancer or inflammation (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY94-9392, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
* Known sensitivity to the study drug or components of the preparation
* Previous treatment with BAY94-9392 in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the accumulation of BAY94-9392 in primary cancer lesions confirmed by histology. | Day 1
Evaluation of the accumulation of BAY94-9392 in known or suspected local and/or systemic recurrent cancer lesions and/or lymph node metastasis or distant metastasis. | Day 1

SECONDARY OUTCOMES:
Standardized uptake value (SUV) | Day 1
Standardized uptake value ratio (SUVR) | Day 1
Vital Signs | Day 1 and Day 2
Laboratory Findings | Day 1 and Day 2
Electrocardiograms (ECGs) | Day 1 and Day 2
Adverse Event Collection | Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Stanford, California, United States

REFERENCES:
- [Derived] Park SY, Na SJ, Kumar M, Mosci C, Wardak M, Koglin N, Bullich S, Mueller A, Berndt M, Stephens AW, Cho YM, Ahn H, Chae SY, Kim HO, Moon DH, Gambhir SS, Mittra ES. Clinical Evaluation of (4S)-4-(3-[18F]Fluoropropyl)-L-glutamate (18F-FSPG) for PET/CT Imaging in Patients with Newly Diagnosed and Recurrent Prostate Cancer. Clin Cancer Res. 2020 Oct 15;26(20):5380-5387. doi: 10.1158/1078-0432.CCR-20-0644. Epub 2020 Jul 21. PMID 32694158
- [Derived] Mittra ES, Koglin N, Mosci C, Kumar M, Hoehne A, Keu KV, Iagaru AH, Mueller A, Berndt M, Bullich S, Friebe M, Schmitt-Willich H, Gekeler V, Fels LM, Bacher-Stier C, Moon DH, Chin FT, Stephens AW, Dinkelborg LM, Gambhir SS. Pilot Preclinical and Clinical Evaluation of (4S)-4-(3-[18F]Fluoropropyl)-L-Glutamate (18F-FSPG) for PET/CT Imaging of Intracranial Malignancies. PLoS One. 2016 Feb 18;11(2):e0148628. doi: 10.1371/journal.pone.0148628. eCollection 2016. PMID 26890637